CLINICAL TRIAL: NCT00620126
Title: The Home Telemanagement (UC HAT) Trial for Patients With Ulcerative Colitis
Acronym: UCHAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: The Broad Foundation (Other); University of Maryland, College Park (Other); Baltimore Research & Education Foundation, Inc. (Other); Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Raymond Cross, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-27882; IBD-0190 (Other Grant/Funding Number: Broad Medical Research Program)
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: Inflammatory bowel disease; Ulcerative colitis; Telemedicine; Telemanagement; Chronic disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): UC Home Automated Telemanagement
  Interventions: Other: UC Home Automated Telemanagement
- Control (Active Comparator): Best Available Care
  Interventions: Other: Best Available Care

INTERVENTIONS:
Other: UC Home Automated Telemanagement — Weekly assessment with UC Home Automated Telemanagement
  Arms: Intervention
Other: Best Available Care — Routine follow up visits and as needed telephone calls and clinic visits, written action plans, educational fact sheets from the CCFA
  Arms: Control

SUMMARY:
The purpose of this study is to determine if home automated telemanagement improves bowel symptoms, quality of life, compliance with medications, and health care utilization compared to best available care in patients with ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a common inflammatory condition of the bowels that results in bloody diarrhea, abdominal pain, and lack of control of bowel movements. UC is a chronic medical condition that causes frequent episodes of symptoms ("flares") followed by symptom-free intervals. Although drugs are available to treat the symptoms, there are obstacles to successful treatment. Because patients need to take medications continuously to avoid flares, compliance with drugs can difficult. Monitoring the symptoms of UC is also challenging, because flares are sporadic and often do not occur at the time of routine office visits. This can result in treatment delays. Although the drugs used to treat colitis are effective, they have side effects which can decrease compliance and quality of life. Patient's knowledge of the disease can also be poor, which can affect many aspects of care.

Telemanagement systems are telemedicine systems that are designed to (1) assist physicians in monitoring their patients, (2) assist physicians in following current guidelines, (3) help patients follow self-care plans, and (4) deliver educational facts to patients. Telemedicine systems have been used in diseases similar to UC and have improved outcomes. We designed a telemanagement system specifically for patients with inflammatory bowel disease (IBD HAT) and found that IBD HAT was easy to use, was accepted by patients, and improved various aspects of patient care including patient knowledge, quality of life, and bowel symptoms.

The purpose of the study is to determine if a home telemanagement system for patients with UC (UC HAT) improves clinical outcomes compared to routine care. Patients with UC will be identified from the University of Maryland IBD program and the gastroenterology clinic of the VA Maryland Health Care System, Baltimore. A computer program will assign interested patients by chance to either the UC HAT or the routine care group. Patients in the UC HAT group will be asked to complete self-testing each week at home using the system. The home-unit consists of a laptop computer and electronic weight scale. After turning on the computer, patients answer questions about their bowel symptoms, medication side effects, and compliance with medications. The home-unit then prompts subjects to measure their weight on the scale. Subjects then receive an educational "tip of the day". The following session, subjects answer an educational question that relates to the tip. After self-testing is completed, the results are transmitted via a phone line to our secure server. The results are made available immediately for review on the physician's web portal. Based on the responses to the symptom diary, side effect questions, medical compliance, and body weight, electronic alerts and action plans can be generated. An alert is sent electronically to the study coordinator, who then reviews the information and discusses the findings with the principal investigator and the patient's medical provider. Changes in patient management can be made if appropriate. An action plan is created for each patient at the first visit and contains a list of tasks for patients to start immediately after self-testing if certain criteria are met. Patients still undergo regularly scheduled clinical visits as prescribed by their medical provider.

Patients assigned to the routine care group will undergo scheduled follow up clinical visits, telephone follow up, and receive educational fact sheets about their disease. This is considered routine care at our centers. All patients will undergo research visits every 3 months for one year. Patients will complete a series of questionnaires at each visit that measure the patient's disease activity, quality of life, IBD knowledge, medical compliance, and other parameters. Emergency room visits and hospitalizations will also be measured. A blood draw is required at each study visit.

We think that UC HAT will improve the monitoring of bowel symptoms and medication side effects and improve medical compliance. These improvements should result in decreased bowel symptoms, improved quality of life, and decreased urgent care visits and hospitalizations. If UC HAT is effective, the system could be used in the IBD community to improve clinical care or be used in patients with limited access to health care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis confirmed by standard clinical, endoscopic, and histologic criteria

Exclusion Criteria:

* Inability to comply with the study protocol
* Previous colectomy with ileostomy or colectomy with ileoanal anastomosis
* History of colonic dysplasia or colorectal cancer
* Uncontrolled medical or psychiatric disease
* Unable or unwilling to provide consent
* Age less than 18 years
* Other forms of colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond K Cross, MD,MS, Principal Investigator — University of Maryland, College Park
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Medical Institute, Baltimore, Maryland

REFERENCES:
- [Background] Cross RK, Arora M, Finkelstein J. Acceptance of telemanagement is high in patients with inflammatory bowel disease. J Clin Gastroenterol. 2006 Mar;40(3):200-8. doi: 10.1097/00004836-200603000-00006. PMID 16633120
- [Background] Cross RK, Finkelstein J. Feasibility and acceptance of a home telemanagement system in patients with inflammatory bowel disease: a 6-month pilot study. Dig Dis Sci. 2007 Feb;52(2):357-64. doi: 10.1007/s10620-006-9523-4. Epub 2007 Jan 9. PMID 17211702

RESULTS

PARTICIPANT FLOW:
Groups:
- UC Home Automated Telemanagement: The UC HAT home unit consists of a netbook computer and an electronic weight scale. Participants answer questions regarding symptoms, side effects, adherence, and receive disease-specific education using the home unit. The home unit automatically transmits the results to the decision support server after each self-testing session. Participants completed self-testing weekly. Updated action plans are automatically transmitted to participant home units if certain criteria are met. If certain clinical conditions are met, email alerts are sent to the nurse coordinator. The coordinator reviews the information and if necessary consults the medical provider and the participant for management changes.
- Best Available Care: The standard of care for participants in this study is modeled after the standard of care at our institution, and based on current evidence-based guidelines including comprehensive assessment, a guideline-concordant therapy plan, scheduled and as needed clinic visits, scheduled and as needed telephone calls, and administration of educational fact sheets about disease-specific topics when appropriate. We expanded the care received by controls to make the groups more comparable. First, we provided the control group with all currently available educational fact sheets from the Crohn's and Colitis Foundation at the time of group allocation. Second, we provided the control group with individualized written action plans at the time of group assignment without reinforcement.
Period: Overall Study
Arm/Group | UC Home Automated Telemanagement | Best Available Care
Started | 25 | 22
Completed | 14 | 17
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (13.9) | 40.3 (13.9) | 41.1 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Clinical Disease Activity (Seo Index)
Description: Clinical disease activity was assessed using the Seo index. An activity index <120 represents clinical remission, whereas scores of 121-150, 151-220, and >221 correlate with mild, moderate, and severe disease respectively. The Seo index is sensitive to change, with a decrease in the index of 35 correlating with a clinical response.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 22
Units | 122 (39.3) | 113.6 (28)

2. Primary Outcome: Quality of Life (IBDQ)
Description: Disease-specific quality of life was assessed using the IBD questionnaire (IBDQ). Scores for the IBDQ range from 32 to 224 with higher scores being associated with better quality of life. Score changes of 16 have been found to be significant changes when compared to baseline values.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 22
Units | 178.1 (32.1) | 187.3 (32.2)

3. Primary Outcome: Percentage of Participants Adherent to Therapy
Description: Adherence was assessed using the Morisky Medication Adherence Score, a 4 item survey in which participants self-report medication-taking behavior. Each question that is answered with a No receives a score of 1. The possible scoring range is therefore 0 to 4. Higher scores correlate with better medical adherence. For the purpose of evaluating percent of participants adherent to therapy, the variable was dichotomized to "Adherent" or "Non-adherent". Any response of Yes to one of the 4 items was scored as "Non-Adherent".
Time Frame: 12 Months
Measure: Number; unit: Percentage of Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 22
Percentage of Participants | 57 | 67

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22

LIMITATIONS AND CAVEATS:
1. Insufficient sample size to detect moderate differences in outcomes between arms
2. Differences between groups at baseline may have resulted in no overall difference between arms at one year
3. Higher rate of attrition than expected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes